CLINICAL TRIAL: NCT04394065
Title: Potential of uEXPLORER Total-body PET/CT in Nasopharyngeal Carcinoma: The Dynamic Imaging, Kinetic Parameters, and Comparison With Conventional PET/CT
Brief Title: uEXPLORER Total-body PET/CT in Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Chief Physician, Sun Yat-sen University
Other Study IDs: 2020-5-13 high-sensitivity PET
Record Dates: First submitted 2020-05-12; First posted 2020-05-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: ultrasensitive PET CT
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- uEXPLORER total-body PET/CT: Newly diagnosed NPC patients will undergo a one-hour total-body dynamic PET/CT examination and subsequently followed by a conventional PET/CT scan within 30 minutes
  Interventions: Device: ultrasensitive positron emission tomography

INTERVENTIONS:
Device: ultrasensitive positron emission tomography — A 194-cm-long total-body positron emission tomography/computed tomography (PET/CT) scanner (uEXPLORER)
  Other Names: conventional PET/CT

SUMMARY:
uEXPLORER total-body PET/CT in Nasopharyngeal Carcinoma

DETAILED DESCRIPTION:
A 194-cm-long total-body positron emission tomography/computed tomography (PET/CT) scanner (uEXPLORER), has been constructed to offer a transformative platform for human radiotracer imaging in clinical research and healthcare. The objective of this study is to determine its specific effect in newly diagnosed nasopharyngeal carcinoma compared with conventional PET/CT and the quantitative kinetic parameters including glucose metabolic rate (Ki), glucose transport rate of flow-in (k1) and flow-out (k2) between tissue and blood, and glucosamine-6-phosphatization rate in tissue (k3). All the neck lymph nodes suspected for metastatic in PET/CT were biopsied under the guidance of ultrasound for a pathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and given written informed consent.
* Aged between 18-65, male/female.
* Histologically confirmed non-keratinizing nasopharyngeal carcinoma (including differentiated type and undifferentiated type, WHO II and III)..
* Fertile women should practice contraception during the study period.
* HGB ≥90g/L ,WBC ≥4*109/L , PLT ≥100*109/L,
* With normal liver function test (ALT and AST ≤2.5*ULN, TBil ≤2.0*ULN)
* With normal renal function test (serum creatinine ≤1.5*ULN)

Exclusion Criteria:

* Women in pregnancy or lactation
* Patients with diabetes
* Prior malignancy except adequately treated basal cell, squamous cell skin cancer, or cervical cancer in situ.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.
* Already involved in other clinical trial.
* Mental disorder, civil disability, limited capacity for civil conduct.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: newly diagnosed NPC
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
The results of uEXPLORER Total-body PET/CT | 6 months
  The Dynamic Imaging, Kinetic Parameters of uEXPLORER Total-body PET/CT

SECONDARY OUTCOMES:
Comparison of uEXPLORER Total-body PET/CT and Conventional PET/CT | 6 months
  Image quality and Static Lesion detectability of TB-PET/CT and conventional PET/CT
Protocol of TB-PET/CT in NPC | 6 months
  Acquisition time and low dose simulation of TB-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, Dr, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Cherry SR, Xie Z, Shi H, Badawi RD, Qi J. Subsecond total-body imaging using ultrasensitive positron emission tomography. Proc Natl Acad Sci U S A. 2020 Feb 4;117(5):2265-2267. doi: 10.1073/pnas.1917379117. Epub 2020 Jan 21. PMID 31964808
- [Result] Lv Y, Lv X, Liu W, Judenhofer MS, Zwingenberger A, Wisner E, Berg E, McKenney S, Leung E, Spencer BA, Cherry SR, Badawi RD. Mini EXPLORER II: a prototype high-sensitivity PET/CT scanner for companion animal whole body and human brain scanning. Phys Med Biol. 2019 Mar 21;64(7):075004. doi: 10.1088/1361-6560/aafc6c. PMID 30620929